CLINICAL TRIAL: NCT03282162
Title: Oxytocin Effects on Neural Processing of Affective Touch and Associations With Trait Autism
Brief Title: The Effects of Oxytocin on Affective Touch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-40
Record Dates: First submitted 2017-09-07; First posted 2017-09-13 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Oxytocin; affective touch; trait autism

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind within-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin then placebo (Experimental): Subjects will first receive oxytocin (24 IU).They then will receive placebo (24 IU) 2 weeks later.
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo
- Placebo then oxytocin (Experimental): Subjects will first receive placebo (24 IU).They then will receive oxytocin (24 IU) 2 weeks later.
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo

INTERVENTIONS:
Drug: intranasal oxytocin — Each subject will be assigned to intranasal administration of oxytocin (24 IU).
Drug: intranasal placebo — An identical amount of intranasal administration of placebo will be assigned to each subject.

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin (24IU) increases the affective processing of touch in general or whether it's effect vary according to the affective valence of the touch (positive, neutral, negative). Moreover, associations with trait autism will be explored.

DETAILED DESCRIPTION:
A double-blind, within-subject, placebo controlled design will be employed in this study. In a randomized-order a total of 40 healthy male subjects will receive oxytocin- and placebo-nasalspray (interval between the administration > 2 weeks). 45 minutes after treatment subjects will be administered the touch-stimulation to the dorsal forearm by a trained experimenter (lengths: 8cm, rate 8cm/s). After each block of stimulation, the subjects will be asked to rate their subjective experience of the touch.The neural basis of touch processing will be measured via simultaneously acquired fMRI.

Levels of trait autism will be assessed using the Autism Spectrum Quotient (ASQ) and related scales such as the Empathy Quotient (EQ), Liebowitz Social Anxiety Scale (LSAS), or the Sensory over Responsivity Scale (SOR) and Under Responsively Scale (URS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury Medical or mental illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
brain function: neural activity during affective touch as assessed via BOLD fMRI | 45-90 minutes after treatment administration
  fMRI data will be analyzed using a within-subject General Linear Model approach - to determine the effects of oxytocin neural activity following oxytocin administration will be compared with neural activity following placebo administration.
Brain function: functional connectivity during affective touch as assessed via BOLD fMRI | 45-90 minutes after treatment administration
  fMRI data will be analyzed using a within-subject General Linear Model approach - to determine the effects of oxytocin on the brain network level, functional connectivity following oxytocin administration will be compared with functional connectivity following placebo administration.

SECONDARY OUTCOMES:
Perceived affective quality of the touch | 45-90 minutes after treatment administration
  Pleasantness ratings of affective touch will be compared between the oxytocin and placebo administration
Associations with trait autism as assessed via the Autism-Spectrum Quotient (AQ) - brain function: activity | 45-90 minutes after treatment administration
  Associations between individual differences in trait autism and brain activity differences between the oxytocin and placebo administration will be examined
Associations with trait autism as assessed via the Autism-Spectrum Quotient (AQ) - brain function: functional connectivity | 45-90 minutes after treatment administration
  Associations between individual differences in trait autism and brain connectivity differences between the oxytocin and placebo administration will be examined
Associations with trait autism as assessed via the Autism-Spectrum Quotient (AQ) - behaviour: pleasantness experience | 45-90 minutes after treatment administration
  Associations between individual differences in trait autism and differences in pleasantness ratings between the oxytocin and placebo administration will be examined
Associations with Sensory Responsivity as assessed via the Sensory Responsivity Scale - brain function: activity | 45-90 minutes after treatment administration
  Associations between individual differences in Sensory Responsivity as assessed via the Sensory Responsivity Scale and brain activity differences between the oxytocin and placebo administration will be examined
Associations with Sensory Responsivity as assessed via the Sensory Responsivity Scale - brain function: functional connectivity | 45-90 minutes after treatment administration
  Associations between individual differences in Sensory Responsivity as assessed via the Sensory Responsivity Scale and brain connectivity differences between the oxytocin and placebo administration will be examined
Associations with Sensory Responsivity as assessed via the Sensory Responsivity Scale - behaviour: pleasantness experience | 45-90 minutes after treatment administration
  Associations between individual differences in Sensory Responsivity as assessed via the Sensory Responsivity Scale and differences in pleasantness ratings between the oxytocin and placebo administration will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Yuanshu Chen, B.S., Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China